CLINICAL TRIAL: NCT05372328
Title: ARMS: The Arm Rest and Support Study
Acronym: ARMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Vital Strategies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB00319633; 139475 (Other Grant/Funding Number: Vital Strategies)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Desk1, Lap, Side, Desk2 (Other): The order of arm positions for participants randomized to this arm will be:
  Desk, Lap, Side, Desk
  Interventions: Other: Position of arm while taking blood pressure measurement
- Desk1, Side, Lap, Desk2 (Other): The order of arm positions for participants randomized to this arm will be:
  Desk, Side, Lap, Desk
  Interventions: Other: Position of arm while taking blood pressure measurement
- Lap, Desk1, Side, Desk2 (Other): The order of arm positions for participants randomized to this arm will be:
  Lap, Desk, Side, Desk
  Interventions: Other: Position of arm while taking blood pressure measurement
- Lap, Side, Desk1, Desk2 (Other): The order of arm positions for participants randomized to this arm will be:
  Lap, Side, Desk, Desk
  Interventions: Other: Position of arm while taking blood pressure measurement
- Side, Lap, Desk1, Desk2 (Other): The order of arm positions for participants randomized to this arm will be:
  Side, Lap, Desk, Desk
  Interventions: Other: Position of arm while taking blood pressure measurement
- Side, Desk1, Lap, Desk2 (Other): The order of arm positions for participants randomized to this arm will be:
  Side, Desk, Lap, Desk
  Interventions: Other: Position of arm while taking blood pressure measurement

INTERVENTIONS:
Other: Position of arm while taking blood pressure measurement — Each participant will have 4 sets of 3 blood pressure measurements taken. The participants will be randomized to the order in which their arm position changes prior to each set of measurements.

SUMMARY:
Primary Objectives

1. Determine the effect of an unsupported and poorly positioned arm on initial and average triplicate blood pressure done according to clinical practice guidelines with an automated device.

a. Hypothesis: Compared to blood pressure measurements obtained with the arm supported with mid-cuff positioned at heart level, blood pressures measured with an unsupported arm and/or with mid-cuff below heart level will be significantly higher.

Secondary Objective

1. To determine if the effects differ based on the following patient characteristics:

* Hypertensive blood pressure (SBP≥130 mmHg vs. <130 mmHg).
* Age (≥ 60 years vs. < 60 years) Greater vascular stiffness > lesser vascular stiffness
* Regular health care (Last BP measured >1 year ago vs. ≤1 year ago)
* Arm length:cuff width

DETAILED DESCRIPTION:
The investigators propose a cross-sectional study of adult participants recruited from the community. Enrolled participants will have four sets of three automated blood pressure measurements, with each set taken with the arm positioned and supported as follows:

* Arm supported on a desk, with mid-cuff at mid-heart level (4th intercostal space)

  * Desk1
  * Reference measurement
* Arm supported on the participant's lap

  * Lap
* Arm hanging at the participant's side, unsupported

  * Side
* The last period of triplicate BP measurements will always have the arm supported and mid-cuff positioned at mid-heart level

  * Desk2

In the prior 3 periods, the arm position and support conditions are randomly ordered. Each participant will undergo a total of 12 systolic and 12 diastolic BP measurements

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Presence of the following on both arms: rashes, gauze dressings, casts, edema, paralysis, tubes, open sores or wounds, A-V shunts.
* Being mentally impaired
* Being pregnant
* Arm circumference exceeding 55 cm.
* >80 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in systolic blood pressure in lap1 vs desk arm position | Time of measurement up to 90 minutes
  Absolute difference between (1) 1st systolic BP and (2) average of 3 systolic BP from measurements (mmHg) obtained in: Lap vs Desk1
Difference in diastolic blood pressure in side vs desk 1 arm position | Time of measurement up to 90 minutes
  Absolute difference between (1) 1st diastolic BP and (2) average of 3 diastolic BP from measurements (mmHg) obtained with: Side vs Desk1
Difference of systolic and diastolic differences | Time of measurement up to 90 minutes
  Systolic and Diastolic BP difference of differences between: (Desk1-Desk2) and (Lap-Desk1) from measurements (mmHg)
Difference of diastolic differences | Time of measurement up to 90 minutes
  Systolic and Diastolic Difference of differences in BP measurements (mmHg) between: (Desk1-Desk2) and (Side-Desk1)

SECONDARY OUTCOMES:
Difference in blood pressure based on hypertension status | Time of measurement up to 90 minutes
  To determine the blood pressure difference based on hypertensive (≥140/90) vs. non-hypertensive participants
Difference in blood pressure based on age | Time of measurement up to 90 minutes
  To determine the blood pressure difference based on age (≥ 60 years vs. <60 years).
Difference in blood pressure based on regular healthcare visits | Time of measurement up to 90 minutes
  To determine the blood pressure difference between participants receiving regular health care visits (>1 year vs. ≤ 1 year).
Difference in blood pressure based on arm length to cuff width ratio | Time of measurement up to 90 minutes
  To determine the blood pressure difference of arm length to cuff width ratio

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Brady, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Liu H, Zhao D, Sabit A, Pathiravasan CH, Ishigami J, Charleston J, Miller ER 3rd, Matsushita K, Appel LJ, Brady TM. Arm Position and Blood Pressure Readings: The ARMS Crossover Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1436-1442. doi: 10.1001/jamainternmed.2024.5213. PMID 39373998